CLINICAL TRIAL: NCT03825094
Title: DyeVert™ System Use for Contrast Monitoring and Minimization in At-Risk Patients Undergoing Angiography Procedures: A Real-World Registry (DyeMINISH Registry)
Brief Title: DyeVert™ System for Contrast Monitoring in At-Risk Patients Undergoing Angiography: A Real-World Registry
Acronym: DyeMINISH
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Osprey Medical, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: TP-6647
Record Dates: First submitted 2019-01-29; First posted 2019-01-31 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Patients at Risk for Developing Contrast-induced Nephropathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: DyeVert™ Contrast Reduction Systems — Osprey Medical DyeVert™ Contrast Reduction Systems (DyeVert Systems) provide fluid pathway resistance modulation such that excess contrast media (CM) (i.e. CM that is not needed for diagnostic or therapeutic purposes) is minimized in the patient's vasculature and total contrast media volume (CMV) reduction occurs, while maintaining adequate image quality.
  Other Names: DyeVert Systems

SUMMARY:
The purpose of this registry-based study is to evaluate the ongoing, real-world clinical performance and safety of commercially available DyeVert Systems during typical clinical use for patients undergoing coronary or peripheral angiography for diagnostic and/or interventional procedures.

DETAILED DESCRIPTION:
Contrast-induced acute kidney injury (CI-AKI) occurs in 3-19% of patients undergoing coronary angiography and is associated with increased morbidity, mortality, and healthcare costs. Patients with chronic kidney disease have greater odds of developing CI-AKI. Guidelines for CI-AKI prevention include screening for risk, volume expansion, and minimizing contrast media volume (CMV) to the patient during angiography; however, hospitals face barriers to implementation in the real-world setting and therefore consistent care delivery for at-risk patients remains a modern clinical challenge. DyeVert Systems provide real-time CMV monitoring and minimization during angiography procedures thereby reducing total CMV to the patient and total CMV relative to baseline renal function, two known risk factors for CI-AKI. The DyeMINISH Registry is designed to evaluate ongoing real-world clinical performance and safety of commercially available DyeVert Systems among a large, real-world population of patients undergoing coronary and peripheral angiography.

ELIGIBILITY:
Inclusion Criteria:

* DyeVert Group Patients: Patient underwent a diagnostic and/or interventional angiography procedure in which the DyeVert System was used in a majority of the case
* Patient is willing and able to provide appropriate informed consent (if required)

Exclusion Criteria:

* Required data was not collected or is not available
* In the Investigator or Sponsor's opinion, the patient is not considered to be suitable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: DyeVert Systems are indicated for patients undergoing angiographic procedures requiring injection of contrast media. Patients at risk for developing contrast-induced nephropathy (CIN) represent the target population for these devices.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2019-05-07 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate contrast media volume (CMV) threshold setting practices and contrast media (CM) usage during index cath lab procedures in which the DyeVert System was used | Index procedure
Evaluate incidence of adverse events associated with index cath lab procedures in which the DyeVert System was used | Index procedure through 120 days post index procedure

CONTACTS AND LOCATIONS:
Overall Officials: Anand Prasad, MD, FACC, Principal Investigator — UT Health Science Center San Antonio: Prof of Medicine & Director Cardiac Catheterization Laboratory
Locations (11):
- United States (11):
  - Hartford Healthcare, Hartford, Connecticut
  - Steward Palmetto General Hospital, Hialeah, Florida
  - Emory Healthcare, Atlanta, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Midwest Heart & Vascular Specialists, Overland Park, Kansas
  - St. Elizabeth Healthcare, Edgewood, Kentucky
  - North Mississippi Medical Center, Tupelo, Mississippi
  - The University of Texas Health Science Center, San Antonio, Texas
  - CHRISTUS Health-Westover Hills, San Antonio, Texas
  - St. Mary's Medical Center, Huntington, West Virginia
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No